CLINICAL TRIAL: NCT03899051
Title: Comparative Clinical Evaluation of Platelet Rich Fibrin and Subepithelial Connective Tissue Graft in Interdental Papilla Reconstruction: A Randomized Controlled Clinical Trial
Brief Title: PRF and Connective Tissue Graft in Interdental Papilla Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: perio isha
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Reconstructive Surgery
Keywords: interdental papilla reconstruction
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Papilla reconstruction would be done with platelet rich fibrin
  Interventions: Procedure: interdental papilla reconstructive surgery with subepithelial connective tissue graft
- Control group (Active Comparator): Papilla reconstruction would be done with subepithelial connective tissue graft
  Interventions: Procedure: interdental papilla reconstructive surgery with PRF

INTERVENTIONS:
Procedure: interdental papilla reconstructive surgery with PRF — Papilla reconstruction would be done with platelet rich fibrin
  Arms: Control group
Procedure: interdental papilla reconstructive surgery with subepithelial connective tissue graft — Papilla reconstruction would be done with subepithelial connective tissue graft
  Arms: Test group

SUMMARY:
Interdental papilla deficiency leads to food impaction, problems with phonetics and an unaesthetic appearance. Reconstruction of the deficient papilla is therefore, important. Perusal of available literature reveals only case reports and case series in the reconstruction of interdental papilla using subepithelial connective tissue graft and platelet rich fibrin autologous graft. Therefore, the current randomized controlled clinical study is intended to compare the effect of platelet rich fibrin and subepithelial connective tissue graft on interdental papilla reconstruction.

DETAILED DESCRIPTION:
INTRODUCTION The rising concern for aesthetics has led to a change in the way dentistry is practised. Modern dentistry, no longer is aimed at only restoration of form and function, but restoration of aesthetics as well. Loss of interdental papilla gives rise to numerous problems such as retention of food, phonetic problems and an unaesthetic look. Reconstruction of this lost interdental papilla is one of the most challenging task as the lack of blood supply is a major obstacle in achieving the desired outcome of any attempts at regeneration.

Subepithelial connective tissue graft has been used for root coverage predictably. Studies in the form of case reports and case series have been done utilizing the connective tissue graft harvested from tuberosity, palate etc with encouraging results in the form of complete or partial interdental papilla fill.

Studies have been done to evaluate the usefulness of platelet rich fibrin(PRF) in regeneration of the interdental papilla. Use of PRF for augmentation of interdental papilla prevents the need for a second surgical site and thereby, the related complications associated with creation of a second surgical site.

On comprehensive search of literature, no study has been evident comparing the effect of subepithelial connective tissue graft and PRF for papilla augmentation. Therefore, the purpose of this study is to compare platelet rich fibrin and subepithelial connective tissue graft in interproximal papilla regeneration. The null hypothesis is that there is no significant difference in the clinical outcome for interdental papilla regeneration by platelet rich fibrin and subepithelial connective tissue graft.

Comparative evaluation of the clinical parameters in interdental papilla reconstruction by using platelet rich fibrin (Test group) and subepithelial connective tissue graft (Control group) MATERIALS AND METHODS The present prospective, analytical, randomized clinical trial will be conducted in the Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences, Rohtak This interventional study includes 36 systemically healthy patients, with class I and class II papillary recession according to Nordland and Tarnow's classification. These will be divided into two groups equally (n = 18) Test group -Papilla reconstruction would be done with platelet rich fibrin Control group -Papilla reconstruction would be done with subepithelial connective tissue graft Patients will be recruited from the outpatient department of Post Graduate Institute of Dental Sciences, Rohtak Single blinding will be adopted where the investigator analysing the results will be unaware to which group the patient belongs.

All the participants will undergo full mouth supragingival and subgingival scaling and root planing with a combination of hand scalers and curettes (Hu Friedy) and ultrasonic scaler (EMS Piezon,250, Switzerland). Oral hygiene instructions will be imparted and will be reinforced at each appointment.

Local anaesthesia in the form of xylocaine HCl (2%) will be administered. 2mm coronal to the mucogingival junction of the involved papilla, a 3-5 mm semilunar incision will be given with an ophthalmic tunnel blade. Crevicular incisions will be given on the necks of the neighbouring teeth on the surfaces adjacent to the papilla defects. Through the semilunar incision given above, free the flap along with papilla from the underlying bone. The tissues will be completely freed from the bone and root, so that coronal displacement of the flap will be possible.

TEST GROUP Platelet rich fibrin (PRF) will be prepared according to the Choukron's protocol.

Trimming of the PRF according to the required size will be done. .PRF will be placed on the recipient site and suturing will be done with a 5-0 vicryl suture.

Periodontal dressing will be given over the surgical area. CONTROL GROUP Subepithelial connective tissue graft will be harvested from the maxillary premolars/first molar region. The graft will be then placed at the recipient site and suturing will be done with 5-0 vicryl suture. Periodontal dressing will be given over the surgical area.

In both the groups post operative instructions will be imparted. Antibiotics and analgesics will be prescribed for 5 days. All patients will be asked to rinse with 0.2% chlorhexidine gluconate twice a day for 2 weeks.

DATA COLLECTION METHODS PPD will be measured using UNC 15 periodontal probe at six sites (mesiobuccal, distobuccal, mesiolingual , distolingual , and median points at buccal and lingual aspect).

GI, PI will be measured using UNC 15 periodontal probe at four sites (distolabial, mesiolabial, labial, lingual gingival margin) Papillary height will be measured from apical aspect of contact point to tip of papilla with UNC 15 probe.

Width of Keratinized Gingiva will be measured with the help of UNC 15 probe from the mucogingival junction to the free gingival margin.

Clinical parameters will be recorded at different time intervals. Healing Index will be measured at 1 week, 2 weeks and 3 weeks. All the other clinical parameters will be measured at baseline, 3 months and 6 months and 1 year. The patients will be reinforced with oral hygiene instructions at every visit.

SAMPLE SIZE CALCULATION Based on data from the previously published study, a difference of 1mm between both test groups (standard deviation: 1.0 mm; significance level alpha: 0.05, power: 0.8) resulted in a sample size of 16 patients . To compensate for possible dropout, 18 patients per group will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age range of 18-55 years who are systemically healthy.
* Patients with class I and class II papillary recession according to Nordland and Tarnow's classification.
* Patients who have completed etiological periodontal therapy (full mouth scaling and root planing) with Plaque index (Silness & Loe) <1, gingival index (Loe & Silness) <1 and showing adequate compliance and willing to participate in the study.

Exclusion Criteria:

* Patients having systemic diseases such as hypertension, diabetes, hyperthyroidism or on medications that influence the outcome of periodontal therapy.
* Presence of open contacts in the maxillary anterior region
* Presence of crowding in the maxillary anterior region.
* Pregnant and lactating women
* Patients with active periodontal disease
* Smokers, tobacco users.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Gain in papillary height | 6 months
  Papillary height will be measured from apical aspect of contact point to tip of papilla with UNC 15 probe.

CONTACTS AND LOCATIONS:
Overall Officials: Nishi Tanwar, MDS, Study Chair — PGIDS,ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India